CLINICAL TRIAL: NCT07370532
Title: Clinical Study to Evaluate Safety and Efficacy of Etoricoxib in Patients With Parkinson's Disease Treated With Conventional Treatment
Brief Title: Etoricoxib in Patients With Parkinsonian Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ihab Elsayed Hassan (Other)
Responsible Party: Sponsor-Investigator, Ihab Elsayed Hassan, Lecturer, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 98658
Record Dates: First submitted 2026-01-17; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Levodopa; Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): (levo-dopa group, n =30) who will receive levo-dopa/carbidopa (125/12.5) mg three times daily for 6 months.
  Interventions: Drug: L-dopa
- Etoricoxib group (Active Comparator): will receive levo-dopa/carbidopa (125/12.5) mg three times daily plus Etoricoxib 90 mg once daily
  Interventions: Drug: L-dopa; Drug: Etoricoxib

INTERVENTIONS:
Drug: L-dopa — Levodopa is the standard therapy in PD.
Drug: Etoricoxib — Etoricoxib, is a selective cyclooxygenase-2 inhibitor. Prostaglandins (PG) are produced from arachidonic acid by the constitutively expressed cyclooxygenase-1(COX-1) and by the inducible COX-2 enzymes and are secreted mainly by astrocytes and microglia.
  Arms: Etoricoxib group

SUMMARY:
Neuroinflammation is considered one of the most important factors contributing critically to pathophysiology of PD . Recently, high mobility group box-1 (HMGB1) protein has been encoded as a potential inflammatory biomarker in PD. HMGB1 mediates immune response mostly through endothelial cells and macrophage activation via targeting two vital cell receptors; Toll-like receptor 4 (TLR4) and advanced glycation end products (RAGE).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Both male and female will be included.
* Patients diagnosed with PD according to Unified Parkinson's Disease Rating Scale.

Exclusion Criteria:

* Breast feeding
* Patients with significant liver and kidney function abnormalities.
* Alcohol and / or drug abusers.
* Patients with known allergy to the study medications
* Pregnant women and women with planned pregnancy.
* Patients who are currently using other anti-inflammatory drugs.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-06-30 (Estimated); Primary Completion 2027-11-10 (Estimated); Study Completion 2027-11-20 (Estimated)

PRIMARY OUTCOMES:
- Change in The Unified Parkinson's Disease Rating Scale | 6 months
  - Change in Unified Parkinson's Disease Rating Scale (UPDRS) Total Score

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt